CLINICAL TRIAL: NCT01009853
Title: A Single Dose, 1-Period, 1-Treatment Study of Codeine Sulfate 15 mg Tablets Under Steady State Conditions
Brief Title: Steady State Study of Codeine Sulfate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CODE-T15-PVFS-1
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O(6)-codeine methyl ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Codeine Sulfate — 15 mg tablet

SUMMARY:
Study to characterize the steady-state pharmacokinetics of codeine and its metabolites morphine, morphine-3-glucuronide (M3G), and morphine-6-glucuronide (M6G) after oral administration of Roxane Laboratories' codeine sulfate tablets administered at a dose of 15 mg Q4H x 5 days.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to codeine sulfate or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick Bieberdorf, MD, Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, Austin, Texas, United States